CLINICAL TRIAL: NCT04574349
Title: Effect of Decompressive Craniectomy Following Traumatic Brain Injury: One Year Study
Brief Title: Decompressive Craniectomy Following Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Eldeen Mohamed Oreaby Adam, Assistant Lecturer at neurosurgery department, Assiut University, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Decompressive craniectomy
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Head Injury Trauma
MeSH Terms: interventions — Decompressive Craniectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Decompressive craniectomy — Removing part of the skull (bone flap) to lower intracranial pressure

SUMMARY:
A prospective clinical trial on trauma patients with increased intracranial pressure(ICP) applied for decompressive craniectomy to lower ICP

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains a major health problem across the globe . Intracranial pressure (ICP) following TBI can be elevated due to increasing mass effect from hematomas, contusions, and diffuse brain swelling. Decompressive craniectomy (DC) is a surgical procedure which involves removing a large part of the skull (bone flap) out to make more room for the swollen brain.Mass lesions can be acute subdural hematoma (ASDH), intraparenchymal, brain oedema, or a combination thereof. The most frequent indication for a DC is an acute subdural hematoma (ASDH). The first modern use of DC following TBI was done by Harvey Cushing in 1908. Cushing treated head-injured patients with a subtemporal DC and he reported a substantial reduction in mortality. The management of TBI progressed significantly in the 21st century due to advances in neuroimaging, prehospital management, neurointensive care, neuroanaesthesia, and rehabilitation. This led to a renaissance of interest in DC for improvement patient conditions. One of the serious concerns regarding DC is that it may reduce mortality, but increase the subset of patients with severe disability and persistent vegetative state. The discrepancy in published outcome may, to some extent, be explained by difference in patient selection, indications, timing , and technique of surgery. In terms of surgical consideration regarding DC, it is now well accepted that the dura mater has to be opened and the minimum diameter of unilateral DC should be around 11-12 cm. Skull reconstruction (cranioplasty) after improvement of neurological state is recommended. Decompressive craniectomy provides additional space for the swollen brain and can effectively reduce ICP, thereby mitigating the risk of herniation. However, despite the positive effect of DC on uncontrollable intracranial hypertension, the effect of surgical decompression in mortality and overall functional outcome following TBI remained controversial.

ELIGIBILITY:
Inclusion Criteria:

* All Patients with signs of increased intracranial tension (subdural hematoma, brain edema, intracerebral hematoma) after trauma diagnosed clinically, radiologically, and resistant to medical decompression.
* Age: up to 60
* Midline shift more than 5 mm.
* GCS > 8

Exclusion Criteria:

* Age: more than 60
* Old trauma
* Unfit for surgery (ex: cardiac patient)
* GCS < 8
* Midline shift less than 5 mm.
* Unwillingness to participate in the study.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of the patient's condition clinically | one year
  Clinically: Change of Glasgow Coma Scale (GCS). Maximum value is 15 Minimum value is 3
Change of the patient's condition radiologically | One year
  By CT brain

CONTACTS AND LOCATIONS:
Overall Officials: Roshdy A Elkhayat, Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] 1. Wilson MH, Kolias AG, Hutchinson PJ. Neurotrauma - a multidisciplinary disease. Int J clic pract 2014;68:5-7. 2. Kolias AG, Kirkpatrick PJ, Hutchinson PJ. Decompressive craniectomy: past, present, and future. Nat Rev Neurol 2013;9:405-15. 3. Sahuquillo J, Arikan F. Decompressive craniecomty for the treatment of refractory high intracranial pressure in traumatic brain injury. Cochrane Database Syst Rev 2010;CD003983. 4. Cushing G. I. subtemporal Decompressive Opertions for the intracranial Complications Associated with Bursting Fractures of the Skull. Ann Surg 1908;47:641-4.1 5. Polin RS, Shaffrey ME, Bogaev, et al. Decompressive bifrontal craniectomy in the treatment of severe refractory posttraumatic cerebral edema. Neurosugery 2015;41:84-92. 6. Whitfield PC, Patel H, Hutchinson PJ, et al. Bifrontal decompressive craniectomy in the management of posttraumatic intracranial hypertension. Br J Neurosurg 2014;15:500-7. 7. De luca GP, Volpin L, Fornezza U, Cervellini P, Zanusso M, Casentini L, Curri D, Piacentino M, Bozzato G, Colombo F, The role of decompressive craniectomy in the treatment of uncontroolable pos-traumatic intracranial hypertension. Acta Neurichir (Suppl) 2000;76:401-404. 8. Faul, F., Erdfelder, E., Lang, A.-G. & Buchner, A. G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behavior Research Methods, 2014;39, 175-191.. 9. I. Timofeev, P.J.Kirkpatrick, E.Corteen, M.Hiller, M.Czosnyka, D.K.Menon, J.D.Pickard, and P.J.Hutchinson Decompressive craniectomy in traumatic brain injury 2006;96:11-16 10. Teasdale G, Jennett B. Assessment of coma and impaired consciousness. Lancet 1974; 81-84 11. Teasdale G, Jennett B. Assessment and prognosis of coma after head injury. Acta Neurochir 1976; 34:45-55.